CLINICAL TRIAL: NCT00647725
Title: Labor Analgesia in the Latent Phrase of the First-stage of Spontaneous Delivery
Brief Title: Labor Analgesia in the Latent Phrase
Acronym: LALP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMU-69714-14XS; MCH03552
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-09

CONDITIONS: Labor Pain
Keywords: Epidural analgesia; Latent analgesia; Active analgesia; Labor delivery
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Active Comparator): Active phrase analgesia
  Interventions: Procedure: Active phrase epidural analgesia
- II (Active Comparator): Latent phrase analgesia
  Interventions: Procedure: Latent phrase epidural analgesia

INTERVENTIONS:
Procedure: Active phrase epidural analgesia — Continuous epidural analgesia with sufentanil plus ropivacaine
  Arms: I
Procedure: Latent phrase epidural analgesia — Continuous epidural analgesia with sufentanil plus ropivacaine
  Arms: II

SUMMARY:
Painless labor is an essential part in woman's health care. Labor analgesia in the active phrase is in popular use currently. However, parturients are still haunted by the labor delivery pain in the latent phrase up to 7-8 hours, especially for the nulliparas. Therefore, we hypothesized that labor analgesia in the latent phrase of the first delivery stage would provide superior health care for laboring women. In addition, such analgesia technique would not prolong the time of uterine dilation and labor delivering.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparas
* Required labor analgesia
* Chinese.

Exclusion Criteria:

* Allergic to opioids and/or local anesthetics
* Failed to performing epidural catheterization
* Organic dysfunction
* Contraindications for epidural analgesia.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15000 (Actual)
Dates: Start 2003-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Rate of Cesarean delivery | The time of the end of the labor

SECONDARY OUTCOMES:
Time of latent phrase | From the beginning of regular contraction of uterus to the diameter of cervix to 4cm
Time of labor | From the beginning of regular contraction of uterus to the end of the labor
Overall feeling of satisfaction of analgesia | From the beginning of regular contraction of uterus to the end of the labor
Side effects | From the beginning of regular contraction of uterus to the end of the labor
VAS pain intensity | From the intinition of analgesia to the cervical dilation >4cm
Instrumental delivery | The end of the time of the labor
Oxytocin infusion rate | During the whole period of laboring
Neonatal Apgar scores | 1st min, 5th min, 10th min and 20th min
Umbilical gas measurement | After delivering of the fetus
Maternal oral temperature | From the initiation of analgesia to the end of the labor
Maternal corticosteroids | 1h before analgesia; 0h of the analgesia; 5min,10min,30min,45min,1h,2h,3h and hourly till the end of the labor

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Result] Wang F, Shen X, Guo X, Peng Y, Gu X; Labor Analgesia Examining Group. Epidural analgesia in the latent phase of labor and the risk of cesarean delivery: a five-year randomized controlled trial. Anesthesiology. 2009 Oct;111(4):871-80. doi: 10.1097/ALN.0b013e3181b55e65. PMID 19741492